CLINICAL TRIAL: NCT00126516
Title: Effects of Angiotensin II Receptor Blockers (ARB) and Angiotensin Converting Enzyme Inhibitors (ACEI) on Progression of Silent Brain Infarction and Cognitive Decline in Japanese Patients With Essential Hypertension in the Elderly
Brief Title: Angiotensin II Receptor Blockers (ARB) and ACE Inhibitors (ACEI) on Silent Brain Infarction and Cognitive Decline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nara Medical University (Other)
Responsible Party: Principal Investigator, Yoshihiko Saito, Professor, Nara Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03-Ken-52
Record Dates: First submitted 2005-08-03; First posted 2005-08-04 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Brain Infarction; Hypertension
Keywords: silent brain infarction; cognitive decline; Angiotensin II Type 1 Receptor Blockers; Angiotensin-Converting Enzyme Inhibitors; hypertension
MeSH Terms: conditions — Brain Infarction; Hypertension; Cognitive Dysfunction | interventions — Angiotensin Receptor Antagonists; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Angiotensin II Receptor Antagonists group
  Interventions: Drug: Angiotensin II Receptor Antagonists
- 2 (Active Comparator): Angiotensin-converting Enzyme Inhibitors group
  Interventions: Drug: Angiotensin-converting Enzyme Inhibitors

INTERVENTIONS:
Drug: Angiotensin II Receptor Antagonists — any dosage, frequency, and duration
  Arms: 1
Drug: Angiotensin-converting Enzyme Inhibitors — any dosage, frequency, and duration
  Arms: 2

SUMMARY:
The purpose of this study is to elucidate whether or not angiotensin II receptor blockers (ARB) are more beneficial or equal to angiotensin converting enzyme inhibitors (ACEI) on development or progression of silent brain infarction and cognitive decline in Japanese patients with essential hypertension in the elderly.

DETAILED DESCRIPTION:
Hypertension plays a major role in the development of cardiovascular diseases. Treating hypertension has been associated with reduction in the risk of stroke and myocardial infarction. Angiotensin converting enzyme inhibitor (ACEI), ramipril, showed a 32 % in relative risk of reduction in the Heart Outcomes Prevention Evaluation (HOPE) trial. Angiotensin II receptor blocker (ARB), losartan, also showed a 25 % in relative risk of reduction in the Losartan Intervention For Endpoint reduction in hypertension study (LIFE).

Elderly people, especially hypertensive patients, with silent brain infarction have an increased risk of stroke and cognitive decline. However, no reports are seen on comparison of the effects of ARBs and ACEIs on progression of silent brain infarction and cognitive decline in patients with essential hypertension in the elderly.

The researchers therefore longitudinally evaluate silent brain infarction using magnetic resonance imaging and cognitive decline by Mini-Mental State Examination twice at an interval of 2 years in patients with essential hypertension in the elderly who are received antihypertensive therapy by ARB or ACEI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension (systolic blood pressure>=140 mmHg and/or diastolic blood pressure>=90, or treated with antihypertensive drugs)
* Patients with any finding of stroke, silent brain infarction, and white matter lesion on magnetic resonance imaging

Exclusion Criteria:

* Secondary hypertension
* Atrial fibrillation
* History or signs of cerebral disorders other than cerebrovascular disease
* Malignant tumor
* Chronic renal failure
* Severe congestive heart failure
* Hyperkalemia
* Stenosis of bilateral renal artery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 395 (Actual)
Dates: Start 2004-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Fatal and nonfatal stroke | two years
Progression of silent brain infarction or white matter lesion on magnetic resonance imaging | two years

SECONDARY OUTCOMES:
Fatal and nonfatal acute coronary syndrome | two years
Admission for heart failure | two years
All cause mortality | two years

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiko Saito, MD, PhD, Principal Investigator — First Department of Internal Medicine, Nara Medical University
Locations (1):
- First Department of Internal Medicine, Nara Medical University, Kashihara, Nara, Japan